CLINICAL TRIAL: NCT05848700
Title: A Double-Blind, Placebo-Controlled, Randomized Withdrawal Study to Evaluate SEP-363856 Physical Dependence in Adult Subjects With Schizophrenia
Brief Title: A Clinical Study to Learn if SEP-363856 Has Physical Dependence in Adults With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEP361-121
Record Dates: First submitted 2023-04-27; First posted 2023-05-08 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856

STUDY DESIGN:
Intervention Model Description: double blind, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SEP-363856 (Experimental)
  Interventions: Drug: SEP-363856
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SEP-363856 — SEP-363856 Tablet
  Arms: SEP-363856
Drug: Placebo — Placebo Tablet
  Arms: Placebo

SUMMARY:
A Clinical Study to learn if SEP-363856 has physical dependence in adults with schizophrenia. This study will be held in approximately 6 study sites in the United States. It will be accepting male and female participants age 18 years to 65 years. Participation will be up to approximately10 weeks.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomized withdrawal study comparing abrupt discontinuation of SEP-363856 (SEP-363856 switched to placebo) to continuous SEP-363856 treatment in male and female adult subjects with schizophrenia.

ELIGIBILITY:
Inclusion Criteria: (this list is not all inclusive)

* Male or female subject between 18 and 65 years of age (inclusive) at the time of informed consent.
* Subject meets Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for a primary diagnosis of schizophrenia as established by clinical interview (using the DSM-5 as a reference and confirmed using the Structured Clinical Interview for DSM-5, Clinical Trials Version [SCID-CT]).
* Subject must have a Clinical Global Impression-Severity Scale (CGI-S) score ≤ 4 (normal to moderately ill) at Screening and Day 1.
* Subject must have a PANSS total score ≤ 80 at Screening and a score of ≤ 4 on the following PANSS items at Screening: P7 (hostility) and G8 (uncooperativeness).
* Subject has been taking an antipsychotic for at least 6 weeks prior to Screening and has had no change in antipsychotic medication(s) (minor dose adjustments for tolerability purposes may be permitted) for at least 6 weeks prior to Screening.

Exclusion Criteria: (this list is not all inclusive)

* Subject has a DSM-5 diagnosis or presence of symptoms consistent with a current DSM-5 diagnosis other than schizophrenia.
* Subject has attempted suicide within 6 months prior to Screening.
* Subject answers "yes" to "Suicidal Ideation" Item 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) on the Columbia Suicide Severity Rating Scale (C-SSRS) at Screening (ie, in the past 1 month) or at any subsequent C-SSRS assessment prior to dosing (ie, since last visit).
* Subject is at significant risk of harming him/herself or others (passive or active) according to the Investigator's judgment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Maximum change from the steady-state baseline (CSSBmax) in the total score of the 20 item Physician Withdrawal Checklist (PWC-20) during the 7-day Randomized Withdrawal Period | up to10 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Woodland International Research Group, LLC, Little Rock, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - Behavioral Clinical Research, Inc, Miami Lakes, Florida
  - Research Centers of America at Fort Lauderdale Behavioral Health Center, Oakland Park, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Neuro-Behavioral Clinical Research, Inc, North Canton, Ohio
  - Pillar Clinical Research, LLC, Richardson, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com